CLINICAL TRIAL: NCT04309721
Title: Efficacy of add-on PEramPanel in Focal Motor Status Epilepticus
Brief Title: Perampanel in Focal Status Epilepticus
Acronym: PEPSI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160949J; 2019-000882-19 (EudraCT Number)
Record Dates: First submitted 2019-12-04; First posted 2020-03-16 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Epilepticus; Status, Focal Motor
Keywords: Perampanel; Placebo; Antiepileptic drug
MeSH Terms: interventions — perampanel; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perampanel (Experimental): immediate enteral administration of Perampanel, 12 mg
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): immediate enteral administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perampanel — Single-dose of Perampanel 12 mg film-coated tablet, will be given orally in patients with status epilepticus that do not involve the oral and pharyngeal musculatures. In alternative, perampanel will be administered by a nasogastric feeding tube, a procedure which has been recently reported to be safe and tolerated in patients with generalised status epilepticus
  Other Names: Experimental group
  Arms: Perampanel
Drug: Placebo — Single-dose of placebo of Perampanel, administered orally. Placebo of perampanel will be given orally, in patients with status epilepticus that do not involve the oral and pharyngeal musculatures. In alternative, Placebo of perampanel will be administered by a nasogastric feeding tube, a procedure which has been recently reported to be safe and tolerated in patients with generalised status epilepticus
  Other Names: Control group
  Arms: Placebo

SUMMARY:
Randomized controlled trial on focal motor status epilepticus (SE), studying the add-on efficacy of the enteral administration of perampanel (PER) to a conventional intravenous antiepileptic drug.

DETAILED DESCRIPTION:
In spite of the use of various antiepileptic drugs, the SE, generalized or focal, are refractory to the treatment in around 25 % of the cases. There is therefore a need to develop new therapy with novel synaptic targets.

New antiepileptic drugs emerge as potential drugs for SE. Perampanel (PER) is a new drug available for add-on therapy in patients with a focal epilepsy. The mechanism of action of this drug is original, as it is a non-competitive α-amino-3-hydroxy-5-methylisoxazole-4-propionate (AMPA) receptor antagonist. Several studies suggested that AMPA-mediated glutamatergic transmission plays an important rule during the SE.

In this study the investigator will focus on patients suffering from early focal motor SE, for several reasons:

(i) There is no randomized controlled double-blind trial in this population, and therefore no evidence to help physicians.

(ii) The investigator aims to perform a trial on early SE, after failure of only one drug (a benzodiazepine, recommended as first line treatment), in order to properly evaluate the effect of the tested drug (add-on of perampanel).

(iii) The perampanel is available only for oral administration. Focal SE usually does not affect the vital prognosis and can be treated less aggressively. Use of oral loading doses of antiepileptic drugs is frequent, and therapies may be changed or adapted in the time-frame of hours or days.

(iv) Patients with a focal SE, presenting motor symptoms, can be included without the need of an EEG. Similarly, the primary end-point, cessation of the motor events, does not require specific exam, and can also be done clinically.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or above, including the protected adults with a focal motor status epilepticus, defined by prominent clinically objective focal motor symptoms (clonic, tonic, myoclonic, adversive or oculoclonic), lasting for more than 10 minutes before any treatment or repeated focal motor seizures during this period (≥ 4 seizures in 10 min)
2. The focal motor status continues (or patients show ≥ 2 focal motor seizures) 5 minutes or more after the beginning of administration of benzodiazepines. The delay between administration of benzodiazepines and randomization must not exceed 6 hours.
3. Affiliation to a French social security system (recipient or assign) excluding "Aide Médicale" Etat (AME)

Exclusion Criteria:

1. Known severe liver (Factor V <50 %) or kidney (glomerular filtration rate : 15-29 ml/min/1,72 m2) insufficiency
2. Women with known or clinically detected pregnancy
3. Patients with known allergies to perampanel or to any of the excipients mentioned in the summary of product characteristics(SmPC)
4. Patients with postanoxic status
5. Patients in coma (Glasgow<8)
6. Patients with motor events for which a nonepileptic psychogenic origin is suspected
7. Patients whose status epilepticus is linked to a pathological condition, such as trauma, who needed immediate surgery
8. Known current treatment by perampanel
9. Known galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption syndrome (rare hereditary diseases)
10. Known participation in another trial with medication and/or previously included in PEPSI study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Administration or not of either (i) an additional second-line antiepileptic drug, either intravenous or orally, or (ii) a third-line (anesthetic drug) | Within de 6 hours after the perampanel or placebo administration
  Administration or not of either (i) an additional second-line antiepileptic drug, either intravenous or orally, or (ii) a third-line (anesthetic drug), within the 6 hours following study drug (perampanel or placebo) administration

SECONDARY OUTCOMES:
Seizure cessation | at 3 hours and 6 hours after the perampanel or placebo administration
  Seizure cessation is defined clinically by the interruption of any epileptic movements (clonic, tonic or myoclonic)
Time to seizure cessation | within the 6 hours after the administration of perampanel or placebo
The need for endotracheal intubation | within the 24 hours after the administration of perampanel or placebo
Percentage of patients with altered consciousness | at 3 hours and 6 hours after the perampanel or placebo administration
  Altered consciousness is defined as Glascow Coma Scale (GCS) <8
Duration of hospitalization | From randomization untill 14 days after the administration of perampanel or placebo
  Duration of overall hospitalization (ICU/step down/standard hospitalisation) and duration of hospitalization in ICU/step down unit, both censored 14 days after randomisation
Rate of patient with seizure recurrence | From hour 3 until hour 24 after the administration of perampanel or placebo
  Seizure recurrence is defined as focal motor seizure lasting less than 10 minutes, between hour 3 and hour 24 after the administration of perampanel or placeb.
  Recurrence is defined by reappearance of epileptic movements after a period of at least one hour of seizure cessation
Rate of patient with status epilepticus recurrence, in patients with seizure cessation | From hour 3 until hour 24 after the administration of perampanel or placebo
  Status epilepticus recurrence is defined as focal motor seizure lasting 10 minutes or more, or repeated focal motor seizures (≥4 seizures in 10 min), between hour 3 and hour 24 after the administration of perampanel or placebo.
Rate of patients with secondary generalized seizures | From hour 0 until hour 24 after the administration of perampanel or placebo
  Secondary generalized seizures is defined as convulsive tonic or clonic bilateral seizure lasting less than 5 minutes
Progression to a convulsive generalized status epilepticus | From hour 0 until hour 24 after the administration of perampanel or placebo
  Convulsive generalized status epilepticus is defined as convulsive tonic or clonic bilateral seizure lasting more than 5 minutes or more, or 2 or more seizures in 5 minutes without recovery of consciousness between the seizures
Mortality rate at the end of the study period | Up to 14 days (end of hospitalization) or 14 days if the patient is still hospitalized
Glasgow Outcome Scale score at the end of the study period | Up to 14 days (end of hospitalization) or 14 days if the patient is still hospitalized
  Glasgow Outcome Scale (GOS) is 5 values score from 1 (death) to 5 (resumption to normal life; there may be minor neurologic and/or psychological deficits).
Global neurological state at the end of the study period | Up to 14 days (end of hospitalization) or 14 days if patient is still hospitalized
  The neurological state of patients will be evaluated for comparison with that before status epilepticus. Three states will be distinguished: unchanged, new neurological deficit or death
Number of adverse events and their severity | from randomization until to 14 days after the administration of perampanel or placebo
Subgroup analysis of the primary and secondary outcomes measure according to the etiology | At H0 (below or above the median of SE duration
  Several etiological categories will be defined :
  * acute symptomatic versus remote symptomatic versus cryptogenic causes
  * identification of a brain lesion versus not
Subgroup analysis of the primary and secondary outcomes measure according to duration of status epilepticus | At H0 (below or above the median of SE duration
Subgroup analysis of the primary and secondary outcomes measure according to type of conventional antiepileptic drug administrated | At H0 (below or above the median of SE duration)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Navarro, DDS,PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (10):
- France (10):
  - Urgences, CHU Lille (Hôpital Roger Salengro), Lille
  - Neuro-physiologie clinique, CHU Lille (Hôpital Roger Salengro), Lille
  - Réanimation polyvalente, CHU (Hopital Roger Salengro), Lille
  - Department of Neurology, Epilepsy Unit, Pitié-Salpêtrière Hospital, Paris
  - Hôpital Pitié Salpêtrière - ICU, Paris
  - Réanimation Polyvalente, GH Paris Saint Joseph, Paris
  - Neurologie et Neurovasculaire, GH Paris Saint Joseph, Paris
  - S.A.U, Pitié-Salpêtrière Hospital, Paris
  - Accueil des Urgences, Centre Hospitalier de Versailles - André Mignot, Versailles
  - Neurologie, Centre Hospitalier de Versailles - André Mignot, Versailles, Île-de-France Region